CLINICAL TRIAL: NCT07116122
Title: A Two-Stage Pilot Study to Evaluate the Feasibility (Stage I) and Efficacy (Stage II) of a Tracking System for Family Caregivers of Persons With Dementia
Brief Title: Evaluating a Wearable Tracking System for Family Caregivers of Persons With Dementia With Wandering Concerns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Koronis Biomedical Technologies (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Colleen Peterson, Assistant Research Scientist, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00241188; 2R42AG058336-02A1 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Memory Loss; Caregiver
Keywords: dementia; memory loss; caregiver; dementia caregiver support; tracking device
MeSH Terms: conditions — Dementia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: A total of 70 (20 in stage 1, 50 in stage II) caregivers as well as the persons with Alzheimer's Disease (AD) will participate. Therefore, the number of anticipated enrollment is 140.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracking/finding system (Experimental): Persons with dementia will wear the tracking device (Care Companion) and the caregivers will be using the companion smartphone application.
  Interventions: Device: Tracking/finding system

INTERVENTIONS:
Device: Tracking/finding system — Persons living with Alzheimer's Disease or Related dementias will wear the Care Companion smartwatch for approximately one month (stage I) or 6 months (stage 2). The Caretakers will utilize the smart phone application (app) to monitor the person wearing the watch and be alerted to elopements. The system will notify a caregiver if the person with dementia leaves a defined area (e.g., the home) via the application. In the tether mode (e.g., outside of the home), the system monitors the distance between the smartwatch and the caregiver's smartphone. When a separation distance exceeds a set threshold, the application will alert the caregiver and start tracking the location of the person with dementia by displaying the person's position on the caregiver's smartphone.

SUMMARY:
This project has two stages feasibility (stage 1) and efficacy of the device (stage II) and is being completed to evaluate a tracking solution system (Care Companion) developed by Koronis Biomedical Technologies (KBT) to assist family caregivers of persons living with dementia that are at risk for wandering/elopement.

Participants in this stage 1 will be involved in this project for approximately 1 month and stage II participants will be involved for approximately 6 months.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Identify as person providing support to the person living with dementia/memory loss due to person's dementia
* Has concerns about person living with dementia/memory loss wandering or eloping
* Have a smartphone (Android or Apple) with sufficient system requirements (e.g., iPhone 4s or better) or indicate a willingness to use the Care Companion and related smart phone application
* Able to converse in English and understand written English
* Must have internet and computer access capable of Zoom
* In the research staff's best judgment can:
* engage and assist the person with dementia wearing the device
* complete surveys via the internet
* engage in feedback on the devices (surveys and, if applicable, interview)

Caregiver Exclusion Criteria:

* Do not meet inclusion criteria
* Are unable to meet device use and orientation schedule requirements

Persons Living with Dementia or Memory Loss Inclusion Criteria:

* Have a provider diagnosis of AD/ADRD or caregiver has demonstrated it via the screening
* Willing to wear the Care Companion device for the duration of the study
* Able to converse in English

Persons Living with Dementia or Memory Loss Exclusion Criteria:

* Do not meet inclusion criteria above
* Currently residing in a nursing home setting without regular outings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Care Companion acceptability and utility (stage I) | 1 Month
  Caregivers will report the utility and perceptions system review checklist with 18 close-ended questions on a 5-point Likert scale (e.g., "Setting up the Care Companion system was easy") and 7 open-ended questions (e.g., "How do think the Care Companion system affected how you care for your relative?"). Scores can range from 18 to 90, with a higher score indicating higher acceptability and utility. Individual items will be reviewed for particular factor utility.
Caregiver Well-Being (stage I) | Baseline and 1 month
  Caregiver burden will be assessed using the 19-item Benjamin Rose Institute Caregiver Strain Instrument. It is rated on a 4-point Likert scale. Scores greater than 8 for Mastery, greater than 10 for Relationship Strain or Health Strain, or greater than 5 for Social Isolation/Activity Restriction may indicate heightened risk and may warrant further clinical investigation.
Wandering and Elopement Behaviors (stage I) | Baseline and 1 month
  Caregivers will use the 27-item Algase Wandering Scale-Version 2 (AWS-V2) measures ambulation patterns to indicate their care recipient's restlessness and inclination to wander and elopement frequency (e.g., boundary transgressions), which has been validated with community-dwelling persons with Alzheimer's Disease Related Dementias (ADRD). This scale will be modified to use the Likert scaling approach to reduce survey burden. The total score ranges from 23-92 with higher scores indicating more frequent wandering behaviors.
Care Companion Semi-Structured Feasibility Interview (stage I) | 1 Month
  All Stage I participants will be asked to participate in a semi-structured interview to learn more about perceptions related cost, sensitivity of the geo-locating, appearance, and privacy or stigma concerns. This information will be summarized into codes and higher level themes using qualitative analysis approaches.
Care Companion acceptability and utility (stage II) | 6 Month
  Caregivers will report the utility and perceptions system review checklist with 18 close-ended questions on a 5-point Likert scale (e.g., "Setting up the Care Companion system was easy") and 7 open-ended questions (e.g., "How do think the Care Companion system affected how you care for your relative?"). Scores can range from 18 to 90, with a higher score indicating higher acceptability and utility. Individual items will be reviewed for particular factor utility.
Caregiver Well-Being (stage II) | Baseline and 6 month
  Caregiver burden will be assessed using the 19-item Benjamin Rose Institute Caregiver Strain Instrument. It is rated on a 4-point Likert scale. Scores greater than 8 for Mastery, greater than 10 for Relationship Strain or Health Strain, or greater than 5 for Social Isolation/Activity Restriction may indicate heightened risk and may warrant further clinical investigation.
Wandering and Elopement Behaviors (stage II) | Baseline and 1 month
  Caregivers will use the 27-item Algase Wandering Scale-Version 2 (AWS-V2) measures ambulation patterns to indicate their care recipient's restlessness and inclination to wander and elopement frequency (e.g., boundary transgressions), which has been validated with community-dwelling persons with Alzheimer's Disease Related Dementias (ADRD). This scale will be modified to use the Likert scaling approach to reduce survey burden. The total score ranges from 23-92 with higher scores indicating more frequent wandering behaviors.
Care Companion Semi-Structured Feasibility Interview (stage II) | 6 Month
  A subset of Stage II participants will be asked to participate in a semi-structured interview to learn more about perceptions related cost, sensitivity of the geo-locating, effect on caregiving, appearance, and privacy or stigma concerns related to the design. This information will be summarized into codes and higher level themes using qualitative analysis approaches.

SECONDARY OUTCOMES:
Alzheimer's Disease (AD) and Alzheimer's Disease Related Dementias (ADRD) Negative Health Events and Service Utilization (stage I) | 1 month
  Number of crises and service utilization (including number of nursing home stays, number of bed days, assisted living stays in the past month, other residential care setting in the past month, overnight hospital stays in past month, and Emergency visits in past month) will be measured with five self-report items. Whether the event happened is a yes/no format, if yes, the study will sum the number of days or events.
Lifespace Questionnaire (stage I) | Baseline and 1 month
  Perceptions of environmental and community mobility of the person with dementia will be assessed with the Lifespace Questionnaire (LSQ). Caregivers will also be asked how frequently the person with dementia took trips outside of the home. The composite score ranges from 0-9, with higher scores representing greater mobility and access to the community and lower scores indicating limited mobility and likely restriction to home.
Alzheimer's Disease (AD) and Alzheimer's Disease Related Dementias (ADRD) Negative Health Events and Service Utilization (stage II) | 6 month
  Number of crises and service utilization (including number of nursing home stays, number of bed days, assisted living stays in the past month, other residential care setting in the past month, overnight hospital stays in past month, and Emergency visits in past month) will be measured with five self-report items. Whether the event happened is a yes/no format, if yes, the study will sum the number of days or events.
Lifespace Questionnaire (stage II) | Baseline and 6 month
  Perceptions of environmental and community mobility of the person with dementia will be assessed with the Lifespace Questionnaire (LSQ). Caregivers will also be asked how frequently the person with dementia took trips outside of the home. The composite score ranges from 0-9, with higher scores representing greater mobility and access to the community and lower scores indicating limited mobility and likely restriction to home.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Peterson, PhD, Principal Investigator — University of Michigan Transportation Research Institute
Locations (1):
- University of Michigan Transportation Research Institute, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No